CLINICAL TRIAL: NCT03151915
Title: Neonatales Outcome Nach Intrauteriner Laserablation Mit 1.0mm-Optik Bei Fetofetalem Transfusionssyndrom
Brief Title: Neonatal Outcome for Laser Coagulation in Twin-to-twin-transfusion Syndrome
Status: Completed | Type: Observational
Sponsor: Michael Tchirikov MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Michael Tchirikov MD, PhD, Professor Dr. med., Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Other Study IDs: NeoTTTS-1
Record Dates: First submitted 2017-05-03; First posted 2017-05-12 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: TTTS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent fetoscopic laser coagulation with TTTS: This is an retrospektive trial. We use data of patients who underwent fetoscopic laser coagulation with TTTS retrospectively. All patients meet eligibility criteria and give written informed consent before therapy. As part of the ongoing quality control we were able to safely store patient data relating to fetoscopic laser coagulation with TTTS.

SUMMARY:
Twin-twin transfusion syndrome is one of the most severe complication in monochorionic twin pregnancies and can cause severe impairment of fetal and neonatal outcome. In severe TTTS the fetoscopic laser coagulation is the treatment of choice. Fetoscopic laser coagulation is associated with a morbidity and mortality due to iatronic rupture of membranes as well as iatrogenic placenta insufficiency. This can cause preterm delivery as well as intrauterine fetal demise. An adaption of the fetoscopic tools to reduce the lesions of the amniotic membrane can decrease the risk of PPROM and increase the overall survival.

DETAILED DESCRIPTION:
Twin-twin transfusion syndrome (TTTS) occurs in approximately 15% of monochorionic pregnancies. The disease is thought to result from unbalanced intertwin blood flow between the donor and the recipient twin through placental vascular anastomoses. Untreated, TTTS is associated with high perinatal mortality and morbidity.

Fetoscopic laser photocoagulation of the vascular anastomoses is currently the best treatment option for TTTS. The aim of laser surgery is to separate completely both fetal circulations by occluding all placental vascular anastomoses.

However, at the same time the fetoscopic procedure can cause injury to the amniotic membrane. This injury will last until childbirth, as the fetal membrane's capability to repair is restricted. This can lead to preterm premature rupture of membranes (PPROM) and in some cases even to fetal loss.

Decreasing the diameter of fetoscopic instruments can reduce injury to the amniotic membrane. At University Hospital Halle/Saale a new ultrathin fetoscpoes with 1.0/1.2 mm optic is used to reduce sheath sectional area from 3.8/4.3 mm (13F) to 2.3mm (7F).

In 2011 the author published a retrospective cohort study of the first results of laser coagulation using 1.0/1.2 mm optic on 27 female patients. The data was compared to the results using 2.0 mm optic on 53 female patients. The comparison brought to light that the survival rate of at least one twin was 97% (compared to 94.4% using classic optic) and 83.3% (75.5%) for both twins surviving. At the same time the use of the ultrathin optic increased the length of pregnancy by 21.3 days, increased the recipient's weight by 389g and also the donor's Apgar score.

On the other hand, donor's weight and recipient's Apgar score remained unchanged. The results also did not show a decrease in the rate of premature rupture of membranes or a decrease in re-TTTS.

The Authors expect to show more advantages using a wider sample size. The data will be analysed adhering to strict quality protocols. This will hopefully allow us to demonstrate our succesful clinical experience with fetoscopic laser photcoagulation for TTTS using a 1.0 mm endoscope.

A retrospective analyse of all data of patients who underwent fetoscopic laser coagulation with TTTS will be performed retrospectively. As part of the ongoing quality control the authors were able to safely store patient data relating to fetoscopic laser coagulation with TTTS. The plan is to compare results using 1.0/1.2 mm optic with 2.0 mm optic.

Planned study areas inlcude gestational age at birth, the child's survival after fetoscopic laser coagulation (at least one child survives, both children survive, intrauterine foetal death of both children), as well as premature rupture of membranes and reoccurrence of TTTS after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of TTTS
* Ability to give informed consent in german or english

Exclusion Criteria:

* Missing informed consent

Ages: 17 Years to 45 Years | Sex: Female
Age Groups: Child, Adult
Study Population: All pregnant women with TTS
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative neonatal survival | 48 hours after fetoscopic surgery
  rate of intrauterine demise until demission
Gestational Age at delivery | at delivery
  average gestational Age at delivery
Long term neonatal survival | fetoscopic surgery until delivery
  rate of fetal demise until delivery

SECONDARY OUTCOMES:
Child's survival after fetoscopic laser coagulation | one minute after delivery
  * at least one child survives
  * both children survive
  * intrauterine foetal death of both children
Premature rupture of membranes | 48 hours after fetoscopic surgery
Reoccurrence of TTTS after the procedure | 48 hours after fetoscopic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Martin-Luther Universität Halle-Wittenberg, Halle, Germany

IPD SHARING:
Plan to Share IPD: Undecided